CLINICAL TRIAL: NCT02348944
Title: Evaluation of Biological Variability in Cartilage Specific Biomarkers (Coll2-1, Coll2-1NO2, FIB3-1 and FIB 3-2) in Healthy Volunteers.
Brief Title: Biological Variability in Cartilage Specific Biomarkers in Healthy Volunteers.
Acronym: COVAR
Status: Completed | Type: Observational
Sponsor: Artialis (Industry)
Responsible Party: Sponsor
Other Study IDs: COVAR
Record Dates: First submitted 2015-01-19; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Effects of; Serum; Urine Marking
Keywords: Biological markers; Cartilage

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Serum and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 15 healthy volunteers: Other: serum and urine sample
  Interventions: Other: serum and urine sample

INTERVENTIONS:
Other: serum and urine sample — Serum and urine samples will be collected at baseline, weeks2, 16, 52 and 68 to assess intra-individual biological variability of cartilage-specific biomarkers Coll2-1/Coll2-1NO2 / FIB3-1 and FIB3-2.

SUMMARY:
The purposes of the study are to assess intra individual biological variability of serum and urinary cartilage specific biomarkers and define the best standardized conditions for blood and urine sampling in the frame of biomarkers dosage.

DETAILED DESCRIPTION:
To assess intra individual biological variability of serum and urinary cartilage specific biomarkers and define the best standardized conditions for blood and urine sampling in the frame of biomarkers dosage. Variation factors assessed are:

* Fasting condition
* Sampling time
* Sampling season
* Physical activity
* Duration and temperature of total blood treatment
* Type of blood collection tube.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged above 18 years.
* Sign an informed consent after being informed
* Able to follow the instructions of the study

Exclusion Criteria:

* Serious associated diseases:

  * Severe liver disease
  * Renal failure
  * HIV
  * hepatitis B or C
* Patient who are the subject of a judicial protection measure or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male or female above 18 years
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Variation of serum and urine sample between baseline, weeks 2, 16, 52 and 68 to assess intra-individual biological variability of cartilage-specific biomarkers Coll2-1/Coll2-1NO2 / FIB3-1 and FIB3-2. | Baseline and weeks 2, 16, 52 and 68
  Change from baseline will be assess by biomarkers dosage using ELISA (Enzyme Linked ImmunoAssay)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Jandrain, MD, Principal Investigator — Clinical Pharmacology Unit, ATC sa, Belgium
Locations (1):
- ATC SA, Unité de pharmacologie clinique, CHU Sart Tilman, Liège, Liege, Belgium